CLINICAL TRIAL: NCT01512134
Title: Deep Brain Stimulation For Morbid, Treatment-Refractory, Obesity
Brief Title: Deep Brain Stimulation for the Treatment of Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Rezai, MD (Other)
Responsible Party: Sponsor-Investigator, Ali Rezai, MD, Professor of Neurological Surgery, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2011H0329
Record Dates: First submitted 2012-01-11; First posted 2012-01-19 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: Obesity; DBS
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBS Surgery (Experimental): All patients enrolled will undergo DBS implantation in the targeted region to assess the safety of the procedure and the efficacy through weight loss.
  Interventions: Device: Deep Brain Stimulation Device

INTERVENTIONS:
Device: Deep Brain Stimulation Device — Deep brain stimulation surgery
  Other Names: Reclaim

SUMMARY:
The purpose of this clinical study is to investigate the safety and efficacy of deep brain stimulation (DBS) as a treatment option for obesity.

DETAILED DESCRIPTION:
The purpose of this clinical study is to investigate the safety and efficacy of deep brain stimulation (DBS) as a treatment option in the management of severe, treatment refractory, morbid obesity.

ELIGIBILITY:
Inclusion Criteria:

* At least 24 months post Roux-en-Y gastric bypass surgery without evidence of a sustained improvement in BMI after gastric bypass surgery for at least 6 months.
* Participant is willing to comply with all follow-up evaluations at the specified times
* Participant is able to provide informed consent
* Fluent in English

Exclusion Criteria:

* Medical contraindications for general anesthesia, craniotomy, or DBS surgery
* Evidence of neurological disorders, e.g., multiple sclerosis, Parkinson's disease and ischemic stroke, or severe brain atrophy or the presence of subdural hygromas or subdural hematomas.
* Severe cardiovascular, pulmonary, renal, liver, hematological disease, severe coagulopathy, acute infectious process

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2012-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Percentage of excess weight loss | 2 years
  The primary outcome measure at the conclusion of the study will be percent of excess weight loss (EWL).

CONTACTS AND LOCATIONS:
Overall Officials: Ali Rezai, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weichart ER, Sederberg PB, Sammartino F, Krishna V, Corrigan JD, Rezai AR. Cognitive Task Performance During Titration Predicts Deep Brain Stimulation Treatment Efficacy: Evidence From a Case Study. Front Psychiatry. 2020 Feb 19;11:30. doi: 10.3389/fpsyt.2020.00030. eCollection 2020. PMID 32140113